CLINICAL TRIAL: NCT05388617
Title: Prospective Clinical Study To Assess The Safety And Efficacy Of A Radiofrequency Diathermocontraction Device For Muscle Stimulation And The Treatment Of Abdominal Fat
Brief Title: Study To Assess Radiofrequency Diathermocontraction Device For Muscle Stimulation And The Treatment Of Abdominal Fat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study stopped because of a business decision.
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED4-PL01-2022
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Muscle Stimulation; Abdominal Fat

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in Group A if they present with abdominal fat and are able to be present for up to 8 treatment visits spaced approximately 1 week apart. Subjects will enroll in Group B for training and experience purposes only and will be able to attend up to 8 treatments spaced at least 3 days apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Experimental): Subjects in Group A will receive up to 8 treatments with the Brera/Med 400 device on their abdomen or flanks. Subjects may receive a phone call 1 week (1-7 days) after each treatment to record side effects. Subjects will return for follow up visits at 30 and 90 days post last treatment for efficacy and side effects assessments.
  Interventions: Device: Brera
- Group B (Experimental): Subjects in Group B may receive up to 8 treatments with the Brera/Med 400 device on their abdomen and/or flanks. Subjects may receive a phone call 1 week (1-7 days) after each treatment to record side effects. Subjects may be asked return for follow up visits at 30 and 90 days post last treatment for efficacy and side effects assessments. Outcome measures will not be taken for subjects enrolled in this group.
  Interventions: Device: Brera

INTERVENTIONS:
Device: Brera — The applicators will be placed in contact with the skin. The entire defined treatment area will then be treated by delivering energy to the skin. Temperature may be continuously monitored and recorded during treatment. Parameters may be adjusted throughout the treatment to increase subject comfort.

SUMMARY:
The intended use of the device in this study to assess the safety and efficacy of the adhesive electrodes for muscle stimulation and the treatment of abdominal fat on the abdomen and/or flanks.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are a healthy male or female 18 years of age or older. Up to 30 subjects will be enrolled at 1 study center. Subjects will be enrolled into 2 groups, Group A and Group B. Subjects will be enrolled in Group A if they present with abdominal fat and are able to be present for all visits as outlined in "Schedule of Visits and Procedures - Group A". Subjects will enroll in Group B for training and experience purposes only and will follow the visit schedule as outlined in "Schedule of Visits and Procedures - Group B".

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 years of age or older.
* Agrees to be treated with the Brera/Med 400 device.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* Is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.
* Has injured (such as a cut, wound) or infected skin, or has presence of evident pathologies such as melanomas or other tumors of the skin, dermatitis, eczema, psoriasis, etc. in the area to be treated.
* Is on local, oral, or systemic anesthetic agents.
* Has nerve insensitivity to heat in the treatment area.
* Has received an organ transplant.
* Has any embedded electronic device that gives or receives a signal, the device should be turned off or removed prior to treatment.
* Has an embedded pacemaker or implantable cardioverter defibrillator (ICD), the client's cardiologist must be consulted prior to treatment.

NOTE: This device has not been tested on patients implanted with electronic devices that receive or emit signals, such as: Pacemakers, Implantable Cardiac Defibrillators (ICD), or Cardiac Resynchronization Therapy (CRT) devices.

* If the neutral pad would need to be placed on a subject that has a metal plate, rod, or any metal implant that could conduct heat.
* Has an allergy to adhesives, such as glues on medical tape, they should be alerted that a rash may occur on the applicator and neutral pad site, and an over-the-counter solution may be used to treat the area.
* Has an unhealthy expectation of the results - this is not plastic surgery and all subjects should be fully informed of the treatment's expected results.
* Has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated - this treatment will be ineffective.
* Has used Accutane (Isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it brittle.
* Is currently taking anticoagulants.
* The treatment area has scars and/or tattoos.
* Has any of the following conditions:

  * Thrombosis or Thrombophlebitis
  * Active Vascular Disease
  * Labyrinthitis and Tinnitus
  * Liver Disease or Dyslipidemias
  * Acute Sepsis
* Has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Cautionary Criteria:

• Has any of the following conditions:

* Autoimmune Disease
* Diabetic
* Herpes Simplex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Director of Clinical Development
Locations (1):
- Cynosure, Inc., Westford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in Group B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 16 | 0 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 0 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 0 | 14
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 0 | 13
  Hispanic | 1 | 0 | 1
  Asian/Indian | 1 | 0 | 1
  Dominican/American | 1 | 0 | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Types range from I-VI, with I meaning little melanin and light hair, and VI representing high amounts of melanin and dark hair. Additional details on this scale can be found in the publication cited for the results section.
  Participants
    Fitzpatrick Skin Type I | 0 | 0 | 0
    Fitzpatrick Skin Type II | 5 | 0 | 5
    Fitzpatrick Skin Type III | 10 | 0 | 10
    Fitzpatrick Skin Type IV | 1 | 0 | 1
    Fitzpatrick Skin Type V | 0 | 0 | 0
    Fitzpatrick Skin Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Satisfied
Description: The number of subjects satisfied with their treatment will be reported.
Time Frame: 30 days follow up.
Population: There were no subjects enrolled for Group B.
Measure: Number; unit: number of participants satisfied
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 0
number of participants satisfied | 10 |

ADVERSE EVENTS:
Time Frame: Adverse events were captured throughout subject participation in the study, approximately 30 days.
Description: 13 out of the 16 subjects who received treatments in Group A observed adverse events.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/0
Other Adverse Events (participants affected / at risk) | 13/16 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=16) | Group B (N=0)
Erythema (Skin and subcutaneous tissue disorders) | 3 | NA
Cramping (Skin and subcutaneous tissue disorders) | 6 | NA
Muscle Twitching (Skin and subcutaneous tissue disorders) | 1 | NA
Pain/Tenderness (Skin and subcutaneous tissue disorders) | 8 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT05388617/Prot_SAP_000.pdf